CLINICAL TRIAL: NCT03630835
Title: 99m Tc-ANNexin-V-128 Scintigraphy for the Identification of Complicated Carotid Atherosclerotic Plaques
Acronym: ANNICA
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Problem of supply of the experimental product (radio tracer).
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P170602; 2017-002952-99 (EudraCT Number)
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Carotid Atherosclerosis; Atherosclerotic Plaque
Keywords: Complicated carotid atherosclerotic plaques; Endarterectomy; 99mTc-ANNexin-V-128
MeSH Terms: conditions — Carotid Artery Diseases; Plaque, Atherosclerotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-Annexin-V-128 uptake on scintigraphy (Experimental)
  Interventions: Other: 99mTc-Annexin-V-128 uptake on scintigraphy

INTERVENTIONS:
Other: 99mTc-Annexin-V-128 uptake on scintigraphy — An intravenous catheter will be placed in the forearm and a dose of 370 Mega-Becquerels of 99mTc-Annexin-V-128 (1-2 ml) over 10 seconds will be injected through the catheter. The patient will wait for 90 minutes in semi-supine position for the clearance of the radiotracer from blood. At 90 minutes p.i., the patient will be placed in a supine position on the bed of a SPECT-CT gamma-camera. A SPECT acquisition including the heart and the brain will be performed over 20 minutes. At the end of the SPECT acquisition, the bed will move to the CT of the imaging system. A CT angiography will be acquired during the intravenous injection of 30-40 ml of iodinated CT contrast agent from the heart to the brain to localize the signal on the SPECT images. The iodinated contrast agent that is currently available at Bichat Hospital for CTA is Iomeron 400 provided by Bracco Imaging.
  The total duration of the imaging study will be 2 hours.

SUMMARY:
The aim of this trial will be to test and validate the value of scintigraphy with injection of 99mTc-Annexin-V-128 for the detection of complicated carotid plaques

DETAILED DESCRIPTION:
Introduction Stroke represents the third cause of death, the first cause of handicap and the second cause of dementia in Europe. Carotid atherosclerotic plaques are the cause of ischemic stroke in about 15 to 20 % of the patients. In presence of carotid stenosis > 50 %, the risk of ischemic stroke is estimated at about 10% per year when the patient has presented symptoms of cerebral ischemia but only at 2% per year in asymptomatic patients. Clinical benefits of surgical carotid endarterectomy have been demonstrated in symptomatic patients with high degree of carotid stenosis, but remain debatable in asymptomatic patients and should be balanced with the risks associated with the revascularization procedure. There is an urgent need to develop imaging tools that improve the identification of patients at highest risk of developing an ischemic stroke Cellular apoptosis is a key feature of ruptured plaques. Apoptotic macrophages release large amounts of tissue factor within the plaque thereby fostering thrombus formation when plaques rupture. Annexin-V is a 36-kDa protein that binds with high affinity and high specificity to phosphatidylserine (PS) head groups expressed on the cell surface at early stages of the apoptotic process. In addition, activated platelets express large amounts of PS at their surface. In a proof-of-concept study, 99mTc-Annexin-V uptake was detected by scintigraphy in carotid atherosclerotic plaques of 4 patients who presented an acute ischemic stroke and was associated with the presence of apoptotic cells on corresponding carotid plaques obtained after carotid endarterectomy procedure.

Design : Monocentric interventional non comparative study Investigational medicinal product(s): 99mTc-Annexin-V-128 Statistical procedure : Statistical analysis will be performed at the end of the study after blinded review and data freezing.

99mTc-Annexin-V-128 uptake will be analyzed as a binary variable considering the presence or absence of detection and as a quantitative variable for the intensity of signal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ Age ≤ 90 years
* Patients with clinical indications to carotid endarterectomy
* Signed the consent form.
* Affiliation of a social security regime

Exclusion Criteria:

* Non-menopausal women
* Chronic kidney disease (eGFR < 45 ml/min/1.73 m2)
* Waldenstrom disease
* Multiple myeloma
* Previous severe adverse reaction to iodinated contrast agent
* Impossibility to stay immobile and maintain the supine position during 20 minutes.
* Altered consciousness or inability to understand the consent form.
* Urinary incontinence without implantation of urinary catheter (risk of urinary contamination).
* Non-atherosclerotic carotid stenosis (history of cervical radiation).
* Patient deprived of liberty or under legal protection measure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
assess the concordance between the detection of 99mTc-Annexin-V-128 uptake on scintigraphy in carotid plaques with SPECT and the presence of complicated plaques on histology obtained after carotid endarterectomy | no later than one month after baseline.
  Concordance will be assessed by Cohen's kappa coefficient between:
  - detection of 99mTc-Annexin-V-128 uptake on scintigraphy in the carotid bulb localized using the CTA 90 minutes after injection of the radiotracer ipsi-lateral to the carotid endarterectomy.
  And
  - presence of complicated atherosclerotic plaques after carotid endarterectomy validated by an Endpoint Adjudication Committee composed of vascular surgeons and pathologists that will review macroscopical aspects of carotid specimen and histology of all explanted carotid plaques.

SECONDARY OUTCOMES:
to evaluate the correlation between the intensity of 99mTc-Annexin-V-128 uptake detected on SPECT and the expression of Annexin-V on immuno-histology of carotid plaques | no later than one month after baseline.
  Correlation: maximal Annexin-V-positive area will be quantified on serial sections of carotid plaques on immunohistochemistry.
to evaluate the relationship between the intensity of 99mTc-Annexin-V-128 uptake detected on SPECT and the morphological aspects of plaques on histology | no later than one month after baseline.
  morphological features of complicated atherosclerotic plaques (thrombus, lipid core, intra-plaque hemorrhage, plaque rupture) detected on histology.
to assess diagnostic performance of 99mTc-Annexin-V-128 scintigraphy for the detection of complicated carotid plaques detected on histology in patients referred for carotid endarterectomy. | no later than one month after baseline.
  Sensitivity and specificity estimation Complicated plaques will be defined as the presence of luminal or intra-plaque thrombus or the presence of plaque rupture detected on the carotid endarterectomy specimen with histology.
to compare the intensity of the 99mTc-Annexin-V-128 uptake in ipsilateral (symptomatic) and contralateral (asymptomatic) carotid artery. | no later than one month after baseline.
  maximal intensity of 99mTc-Annexin-V-128 uptake on scintigraphy in the carotid bulb localized using the CTA 90 minutes after injection of the radiotracer contralateral to carotid endarterectomy.
to test the intra- and inter-operator reproducibility of the analysis of 99mTc-Annexin-V-128 uptake in carotid bulb | no later than one month after baseline.
  Intra class correlation coefficients between operator measurement as Research methodology

CONTACTS AND LOCATIONS:
Overall Officials: Pierre AMARENCO, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No